CLINICAL TRIAL: NCT05965336
Title: Walking Function in Individuals With Diabetic Peripheral Neuropathy: Biomechanical Mechanisms and Implications for Clinical Outcomes and Gait Retraining
Brief Title: Walking Function in Diabetic Peripheral Neuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Institute for Human and Machine Cognition (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Nicole Rendos, Research Scientist, Florida Institute for Human and Machine Cognition
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-2025-0002; K01HD107294 (NIH)
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetes; Biofeedback-induced changes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: To evaluate biofeedback-induced changes in plantar pressure, propulsion, and biomechanics during gait in individuals with DPN versus age-similar controls. Then, participants with DPN will will complete an additional four experimental sessions to collect data in a randomized crossover pilot clinical trial to examine the acceptability, feasibility, safety, and preliminary effects of gait biofeedback training in individuals with DPN.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Able-Bodied Participants (Active Comparator): Able-bodied participants will complete a total of three study sessions. The three sessions include a clinical evaluation, gait biomechanics, and gait biofeedback for comparison with participants with DPN.
  Interventions: Other: Clinical Evaluation; Other: Evaluation of Passive Ankle Stiffness; Other: Gait Biomechanics; Other: Gait Biofeedback
- Plantar Pressure Biofeedback Gait Training Followed by Propulsion Biofeedback Gait Training (Experimental): Participants with DPN will complete a total of seven study sessions. The first three sessions include a clinical evaluation, gait biomechanics, and gait biofeedback for comparison with able bodied participants. Sessions four through seven involve two different biofeedback training sessions followed by a retention gait analysis test 24-48 hours after training. Participants in this study are are randomized to receive plantar pressure biofeedback gait training first and propulsion biofeedback gait training at least three weeks later.
  Interventions: Other: Clinical Evaluation; Other: Evaluation of Passive Ankle Stiffness; Other: Gait Biomechanics; Other: Gait Biofeedback; Other: Plantar Pressure Biofeedback Gait Training; Other: Propulsion Biofeedback Gait Training
- Propulsion Biofeedback Gait Training Followed by Plantar Pressure Biofeedback Gait Training (Experimental): Participants with DPN will complete a total of seven study sessions. The first three sessions include a clinical evaluation, gait biomechanics, and gait biofeedback for comparison with able bodied participants. Sessions four through seven involve two different biofeedback training sessions followed by a retention gait analysis test 24-48 hours after training. Participants in this study are are randomized to receive propulsion biofeedback gait training first and plantar pressure biofeedback gait training at least three weeks later.
  Interventions: Other: Clinical Evaluation; Other: Evaluation of Passive Ankle Stiffness; Other: Gait Biomechanics; Other: Gait Biofeedback; Other: Plantar Pressure Biofeedback Gait Training; Other: Propulsion Biofeedback Gait Training

INTERVENTIONS:
Other: Clinical Evaluation — A clinical evaluation occurs at the first study session. The clinical evaluation assesses walking function and mobility, lower extremity, sensation, health-related quality of life (HRQoL) and foot function.
  Session 2 will be a dynamometer-based evaluation of passive ankle stiffness and 3-dimensional gait analysis to evaluate baseline biomechanics. During Session 3, real-time biofeedback conditions will be used to measure the immediate effects on walking function.
Other: Evaluation of Passive Ankle Stiffness — Participants will be seated in a dynamometer with their trunk and thigh stabilized to the dynamometer chair, ankle joint aligned with the rotational axis of the dynamometer, and foot stabilized to the foot plate. EMG activity will be recorded from lower limb muscles (gastrocnemius, soleus, tibialis anterior) during all isolated contractions. Participants will first perform three maximum voluntary isometric contractions (MVIC) while seated in a dynamometer. Participants will then perform three isokinetic dorsiflexion tasks while using electromyographic biofeedback at a prescribed level of 50% MVIC soleus activation. The slope of the linear best fit line from the ankle moment vs. angle plot will yield total ankle joint stiffness (i.e., active + passive) at a fixed activation. In three additional trials, the dynamometer will move the ankle joint through the same motion without active subject resistance and the same analytical procedures will derive passive ankle joint stiffness.
Other: Gait Biomechanics — Three-dimensional gait analysis is performed as participants walk at a self-selected speed on an instrumented treadmill. Reflective markers are attached to lower extremity segments. Elastic bands are wrapped around the thighs, calves, and pelvis to which small, thermoplastic shells containing reflective markers are attached. Additional markers are taped to the participant's shoes and on the upper back, shoulder, hip, knee, and ankle joints with adhesive skin tape. Marker data is collected using a 7-camera motion analysis system (Vicon Inc., USA). Vicon motion analysis cameras will collect the location of the retroreflective markers in Vicon Nexus software.
Other: Gait Biofeedback — Audio-visual biofeedback will be provided using a screen placed in front of the treadmill and a speaker. For plantar pressure biofeedback, a visual display of a foot with a colored heat map will represent the current plantar pressure, in addition to bar graphs representing real-time movement of plantar pressure in specific areas of the foot. A target will be provided using the heat map colors of red and target line on the bar graph. For propulsion biofeedback, a visual display with a marker will represent the current propulsion (peak AGRF) and a target provided to modulate propulsion. The plantar pressure and AGRF measurements from the participant's baseline walking trials will be used to determine customized biofeedback targets.
Other: Plantar Pressure Biofeedback Gait Training — Participants will complete a 3-dimensional gait evaluation prior to training, after a 6-minute control bout without biofeedback, and following three 6-minute biofeedback training bouts (total 18-minutes). Individualized biofeedback targets will be calculated from each participant's immediate biofeedback session to best minimize plantar pressure whilst maintaining or enhancing propulsion. Audio-visual biofeedback is provided using a screen placed in front of the treadmill and a speaker. For plantar pressure biofeedback, a visual display of a foot with a colored heat map represents the current plantar pressure, in addition to bar graphs representing real-time movement of plantar pressure in specific areas of the foot. A target is provided using the heat map colors of red and target line on the bar graph. Participants are informed that the target is a measurement of the pressure under their foot, and their goal is to decrease pressure to achieve their target.
  Arms: Plantar Pressure Biofeedback Gait Training Followed by Propulsion Biofeedback Gait Training; Propulsion Biofeedback Gait Training Followed by Plantar Pressure Biofeedback Gait Training
Other: Propulsion Biofeedback Gait Training — Participants will complete a 3-dimensional gait evaluation prior to training, after a 6-minute control bout without biofeedback, and following three 6-minute biofeedback training bouts (total 18-minutes). Individualized biofeedback targets will be calculated from each participant's immediate biofeedback session to best minimize plantar pressure whilst maintaining or enhancing propulsion. Audio-visual biofeedback is provided using a screen placed in front of the treadmill and a speaker. For propulsion biofeedback, a visual display with a marker represents the current propulsion (peak AGRF) and a target provided to modulate propulsion. Participants are informed that the marker is a measurement of how hard they are pushing the ground backward, and their goal is to push-off more to achieve their target.
  Arms: Plantar Pressure Biofeedback Gait Training Followed by Propulsion Biofeedback Gait Training; Propulsion Biofeedback Gait Training Followed by Plantar Pressure Biofeedback Gait Training

SUMMARY:
The purpose of this study is to 1) examine the differences in walking function and movement patterns between individuals with diabetic peripheral neuropathy and healthy adults with no known conditions; 2) examine if receiving feedback on walking form will help change walking patterns; and 3) examine the feasibility, safety, and preliminary effects of walking training with feedback on walking function in individuals with diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
Over 34 million adults in the United States are living with Diabetes Mellitus (DM). Diabetic peripheral neuropathy (DPN) is the most common complication, affecting 50% of individuals with DM. Consequences of DPN include reduced sensation and feedback from the foot and lower limb and increased plantar pressures, predisposing patients to ulcers and lower extremity amputation. Individuals with DPN experience decreased quality of life compared with their healthy and non-neuropathic DM peers, and report problems with mobility, daily activities, pain, and discomfort. Additionally, people with DPN display reduced functional ambulation, step counts, and walking speed. Though increases in physical activity and functional capacity have been associated with improvements in quality of life, DPN poses a unique challenge in mitigating risk while pursuing traditional exercise and walking programs.

Traditional gait training programs used to improve walking function may increase ulceration risk, making these interventions unsuitable if not tailored for people with DPN. The goal of this study is to elucidate the underlying biomechanical mechanisms contributing to the inter-relationships between plantar pressure and propulsion in individuals with DPN, and to examine the safety and feasibility of using real-time biofeedback to modify plantar pressure and propulsion during gait.

The aims of this study are to evaluate (1) biomechanical mechanisms contributing to abnormal plantar pressure and propulsion during gait in individuals with DPN; (2) biofeedback-induced changes in plantar pressure, propulsion, and biomechanics during gait in individuals with DPN and age-similar controls; and (3) the acceptability, feasibility, safety, and preliminary effects of gait training in individuals with DPN. Insights into the biomechanical mechanisms underlying plantar pressure and propulsion in people with DPN will allow for the design of more informed and effective gait rehabilitation interventions aimed at preventing deleterious outcomes such as ulceration and amputation that can be tailored to individual patient characteristics.

Able-bodied participants will complete three experimental sessions and participants with DPN will complete a total of seven experimental sessions. Each session will be approximately 2-3 hours in duration.

ELIGIBILITY:
Inclusion Criteria for All Participants:

1. Age 45+ years
2. Able to walk 10-meters independently without an assistive device
3. Sufficient cardiovascular and musculoskeletal health to walk on a treadmill for 1-minute at self-selected speed

Inclusion Criteria for Participants with DPN:

1. Diagnosis of DM
2. Diagnosis of DPN by a physician
3. Foot examination within the past 6 months to document ambulatory status
4. Physician's clearance

Exclusion Criteria for Healthy Able-Bodied Individuals:

1. History of neurologic disease
2. History of orthopaedic disease affecting the lower extremities
3. History of injury or pain affecting the lower extremity or walking function within the past 6 months

Exclusion Criteria for All Participants:

1. History of amputation
2. Active ulceration
3. Medial column deformity
4. History of Charcot osteoarthropathy
5. History of posterior muscle group lengthening
6. History of lower extremity joint replacement
7. History of lower extremity and/or foot surgery affecting walking mechanics
8. Orthopaedic problems of the lower limbs or spine due to other medical conditions (not DM or DPN) that limit walking or cause pain during walking
9. Improper footwear for walking and community ambulation
10. Cardiovascular or medical condition affecting ability to walk safely
11. History of unexplained dizziness or fainting in the past 2 months
12. Allergy to adhesive tape or rubbing alcohol
13. Individuals who are pregnant, prisoners, or not yet adults
14. Inability to communicate with the investigators
15. Inability to provide written informed consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Biomechanical plantar pressure | Study Session 2 (occurs 24 hours up to 2 weeks after Day 1)
  Plantar pressure is calculated in kilopascals (kPa) using a force sensor placed between the participant's foot and insole of their shoe. The peak plantar pressure in regions of interest (forefoot) will be calculated.
Biomechanical Propulsion | Study Session 2 (occurs 24 hours up to 2 weeks after Day 1)
  Propulsion is calculated as the maximum anteriorly directed ground reaction force during the stance phase of gait using the instrumented (force plate) treadmill.
Biomechanical modulation of ankle stiffness | Study Session 2 (occurs 24 hours up to 2 weeks after Day 1)
  Participants will walk for 3 minutes on a treadmill at their self-selected speed to enable stabilization of movement patterns, warmup, and preconditioning of lower extremity muscles prior to dynamometer tasks. Participants will then be seated in a dynamometer with their trunk and thigh stabilized to the dynamometer chair, ankle joint aligned with the rotational axis of the dynamometer, and foot stabilized to the foot plate. Electromyography (EMG) activity will be recorded from lower limb muscles during all isolated contractions. Participants will first perform three maximum voluntary isometric contractions (MVIC) while seated in a dynamometer. Participants will then perform three isokinetic dorsiflexion tasks while using electromyographic biofeedback at a prescribed level of 50% MVIC soleus activation. The slope of the linear best fit line from the ankle moment vs. angle plot will yield total ankle joint stiffness at a fixed activation.

SECONDARY OUTCOMES:
Changes induced by biofeedback in plantar pressure | Study sessions 4 (48 hours - 3 weeks after session 3), 5 (24-48 hours after session 4) , 6 (3 weeks after session 5) and 7 (24-48 hours after session 6)
  Plantar pressure measurements will be recorded using insoles placed between the surface of the foot and the insole of the participant's shoe. Marker data, GRFs, and plantar pressure data will be synchronized.
  Regression analysis will be used to examine plantar pressure during gait by study group.
Changes induced by biofeedback in propulsion | Study sessions 4 (48 hours - 3 weeks after session 3), 5 (24-48 hours after session 4) , 6 (3 weeks after session 5) and 7 (24-48 hours after session 6)
  Ground reaction force (GRF) data will be collected independently from each leg using a split-belt treadmill instrumented with two 6-degree of freedom force platforms. The antero-posterior GRFs (AGRF) will be used to compute propulsion.
  Regression analysis will be used to examine propulsion during gait by study group.
Changes induced by biofeedback in biomechanics during gait | Study sessions 4 (48 hours - 3 weeks after session 3), 5 (24-48 hours after session 4) , 6 (3 weeks after session 5) and 7 (24-48 hours after session 6)
  Lower extremity kinetics and kinematics will be measured using a three-dimensional motion analysis system and split-belt instrumented treadmill. Kinetics and kinematics of the ankle, knee, and hip will be analyzed during gait.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Rendos, PhD, Principal Investigator — Research Scientist
Locations (1):
- Florida Institute for Human and Machine Cognition, Pensacola, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie published results will be made available for sharing with other researchers after de-identification.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 12 months and ending 36 months following publication of the the findings from this study.
Access Criteria: Data will be available to be shared with scientific and clinical collaborators, clinical and research communities, for individual participant data meta-analyses. Requests should be directed to nrendos@emory.edu and may be submitted up to 36 months following publication of this study. To gain access, data requestors will need to sign a data access agreement.